CLINICAL TRIAL: NCT06017635
Title: Non-invasive Monitoring and Serum Marker Study in Children With Cerebral Edema
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202306-010
Record Dates: First submitted 2023-08-01; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-07

CONDITIONS: Brain Edema
MeSH Terms: conditions — Brain Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: 1. Age 1-18 years old, male or female. 2. Diagnosed with cerebral contusion/cerebral hemorrhage/intracranial tumor postoperative / intracranial infection/septic encephalopathy/metabolic encephalopathy. 3. The research purpose, significance, risks, benefits, and informed consent of patients and their families to the study.
  Interventions: Other: Exposure factors
- Contral: 1. Age 1-18 years old, male or female. 2. Non-cranial organic injury diseases. 3. Physical condition allows them to participate in the study. 4. The research purpose, significance, risks, benefits, and informed consent of patients and their families to the study.
  Interventions: Other: Exposure factors

INTERVENTIONS:
Other: Exposure factors — 1. General information Name, gender, age, weight (kg), major diseases
  2. Clinical data:
  Non-contrast CT scan results of cranial CT on the first day of admission, serum SUR1, trpm4 and MMP-9 expression on the 1st, 4th, 7th and 14th days of admission, S100-β and NSE values on the 1st, 4th, 7th, and 14th days of admission, disturbance coefficient on the 1st, 4th, 7th, and 14th days of admission, Glasgow coma score on the 1st, 4th, 7th, and 14th days of admission, GOS-E score and Merriam-Webster Intelligence Scale score at 3 months of discharge.

SUMMARY:
Purpose of the study：This study aimed to evaluate the clinical significance of serum SUR1, TRPM4 and MMP-9 in the diagnosis of cerebral edema in children with cerebral edema admitted to PICU by comparing them with CT results and perturbation coefficients, so as to provide biological indicators for clinical diagnosis of cerebral edema and provide targets for the treatment of cerebral edema in various diseases.

DETAILED DESCRIPTION:
Early and efficient use of various measures to control and monitor peripheral cerebral edema and intracranial pressure, timely and accurate adjustment of treatment plan to reduce the degree of cerebral edema and reduce intracranial pressure, can significantly improve the development of the disease and prognosis recovery. At present, the clinical diagnosis of cerebral edema is mainly through clinical manifestations and imaging examinations, and there is a lack of corresponding biological examination methods.Purpose of the study：1.By analyzing the correlation between serum SUR1, TRPM4, MMP-9 and the electromagnetic disturbance coefficient, cranial CT results, Glasgow coma score, S100-β, NSE and prognostic score at 3 months of discharge, the clinical value of serum SUR1, TRPM4, MMP-9 and perturbation coefficient in the diagnosis, intracranial pressure monitoring, condition assessment and prognosis judgment of cerebral edema in children was explored.2.By analyzing the changes of the above indicators in various children with cerebral edema admitted to PICU, the types of cerebral edema and the cellular and molecular mechanisms of cerebral edema caused by different diseases were explored.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-18 years old, male or female
* Diagnosed with cerebral contusion/cerebral hemorrhage/intracranial tumor postoperative / intracranial infection/septic encephalopathy/metabolic encephalopathy.
* The research purpose, significance, risks, benefits, and informed consent of patients and their families to the study.

Exclusion Criteria:

* Critically ill and not suitable for research.
* Those who are allergic to electrode sheets and do not cooperate.
* Age> 18 years old or < 1 month.
* Failure to obtain written permission from the guardian.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children whose PICU income meets the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Serum SUR1 concentration | On days 1, 4, 7, and 14 of enrollment
Serum TRPM4 concentration | On days 1, 4, 7, and 14 of enrollment
Serum MMP-9 concentration | On days 1, 4, 7, and 14 of enrollment
Perturbation coefficient monitored by noninvasive cerebral edema monitor | On days 1, 4, 7, and 14 of enrollment
Area of cerebral edema as shown on cranial CT | Day 1 of admission

CONTACTS AND LOCATIONS:
Overall Officials: XinJie Liu, Study Director — Director of Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No